CLINICAL TRIAL: NCT07232628
Title: Energy Availability in Elite Triathletes: Impact on Performance and Injury Risk
Brief Title: Energy Availability and Its Impact in Elite Triathletes
Acronym: TriatLEA
Status: Recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jakob Agergaard, Senior Researcher, Ph.D., Bispebjerg Hospital
Other Study IDs: BBH171; H-25043062 (Other: The Regional Health Research Ethics Committees for the Capital Region of Denmark)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Low Energy Availability; Relative Energy Deficiency in Sport
Keywords: RED-S; injury risk; performance; triathlon; biomarker
MeSH Terms: conditions — Relative Energy Deficiency in Sport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Triathletes: Elite triathletes

SUMMARY:
This study investigates how energy availability affects performance, injury risk, and training outcomes in elite triathletes. Over two competitive seasons (2026-2027), 40 elite and sub-elite triathletes will be monitored through physiological tests, blood samples, and questionnaires. The goal is to identify markers of low energy availability and understand its impact on health and athletic performance. The study is observational and does not involve experimental treatments. Participants continue their regular training and diet while undergoing periodic assessments.

DETAILED DESCRIPTION:
Low energy availability (LEA) is a condition where the energy intake of an athlete is insufficient to support both training demands and essential physiological functions. LEA is common among endurance athletes, including triathletes, due to high training volumes and sometimes intentional dietary restrictions. Prolonged LEA can lead to hormonal imbalances, impaired bone health, reduced immune function, and increased injury risk. This study aims to explore the prevalence and consequences of LEA in elite triathletes over two seasons.

The study is a 2-year exploratory cohort study conducted at the Institute of Sports Medicine, Bispebjerg Hospital, Copenhagen. Forty elite or sub-elite triathletes (men and women, aged 18+) who train more than 15 hours per week will be enrolled. Participants will undergo five comprehensive test days spaced across the off-season, pre-season, and in-season periods of 2025-2027. These test days include blood sampling, DXA scans, MR imaging, muscle strength and stiffness assessments, VO₂ max testing, and dietary and activity monitoring.

The primary outcome is the change in the thyroid hormone triiodothyronine (T3), a known marker of LEA. Secondary outcomes include bone density, muscle mass, metabolic rate, performance metrics (e.g., running economy, VO₂ max), and injury incidence. Energy availability will be assessed via validated questionnaires (LEAF-Q for females, LEAM-Q for males), dietary logs (MyFood24), and training data from wearable devices.

Monthly injury reports and quarterly dietary assessments will be collected. Blood samples will be analyzed for hormones (e.g., cortisol, testosterone, GH, IGF-1, TSH, T3, T4), bone turnover markers (CTX, PINP, osteocalcin), immune parameters, and nutritional status (e.g., vitamin D, iron, B12). Some samples will be stored in a coded biobank until 2029 for future analysis.

Participants will receive no financial compensation but will be reimbursed for public transport. All procedures are non-invasive or minimally invasive and carry low risk. The study has been approved by the relevant ethics committee (Approval No. H-25043062), and informed consent will be obtained from all participants.

Results will be published in peer-reviewed journals and presented at scientific conferences. If not accepted for publication, results will be made publicly available via ClinicalTrials.gov and the EU Clinical Trials Register.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Healthy individuals
* Training ≥15 hours/week in triathlon

Exclusion Criteria:

* Smokers
* Use of prohibited substances (WADA list) without medical justification
* Existing injuries or illnesses that could worsen due to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elite triathletes with a weekly training volume of more than 15 hours
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
T3 | Two years - from off-season 2025 until in-season 2027
  Plasma triiodothyronine (T3) levels

SECONDARY OUTCOMES:
RER | Two years - from off-season 2025 until in-season 2027
  Resting energy expenditure by indirect calorimetry
Bone mineral density | Two years - from off-season 2025 until in-season 2027
  Bone mineral density by DXA scanning
Fat free mass | Two years - from off-season 2025 until in-season 2027
  Fat free mass by DXA scanning
Appendicular fat free mass | Two years - from off-season 2025 until in-season 2027
  Appendicular fat free mass by DXA scanning
Fat mass | Two years - from off-season 2025 until in-season 2027
  Fat mass by DXA scanning
Tendon thickness | Two years - from off-season 2025 until in-season 2027
  Patella and Achilles tendon thickness by ultrasound
Tendon vascularisation | Two years - from off-season 2025 until in-season 2027
  Color doppler by ultrasound of Patella and Achilles tendons
Tendon stiffness | Two years - from off-season 2025 until in-season 2027
  Patella and Achilles tendon stiffness by MyotonPro measurement
Quadriceps muscle strength | Two years - from off-season 2025 until in-season 2027
  Concentric muscle strength by Biodex dynamometer
Hamstring muscle strength | Two years - from off-season 2025 until in-season 2027
  Concentric muscle strength by Biodex dynamometer
Peak muscle power | Two years - from off-season 2025 until in-season 2027
  Measured during counter movement jump on force-plate
Jump height | Two years - from off-season 2025 until in-season 2027
  Measured during counter movement jump on force-plate
Running economy | Two years - from off-season 2025 until in-season 2027
  Measured on treadmill with direct measurement of oxygen uptake
Biking economy | Two years - from off-season 2025 until in-season 2027
  Measured on ergometer bike with direct measurement of oxygen uptake
Maximal oxygen uptake | Two years - from off-season 2025 until in-season 2027
  Measured on ergometer bike with direct measurement of oxygen uptake
Calorie intake | Two years - from off-season 2025 until in-season 2027
  Measured on three-day dietary registrations
Exercise energy expenditure | Two years - from off-season 2025 until in-season 2027
  Measured by tracking devices
Risk of low energy availability | Two years - from off-season 2025 until in-season 2027
  Evaluated by questionnaires - LEAF-Q for females, and LEAM-Q for males
Risk of eating disorder | Two years - from off-season 2025 until in-season 2027
  Evaluated by EDE-Q questionnaire
Injury prevalence | Two years - from off-season 2025 until in-season 2027
  Evaluated through monthly injury diary
Time loss due to injuries | Two years - from off-season 2025 until in-season 2027
  Evaluated through monthly injury diary
Biomarkers | Two years - from off-season 2025 until in-season 2027
  Biomarkers related to metabolism, stress hormones, sex hormones, immune system, muscle breakdown, organ function, bone turnover, lipid profile, minerals, haemoglobin and iron status measured from blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.bispebjerghospital.dk/afdelinger-og-klinikker/institut-for-idraetsmedicin/forskning/Sider/Triatleter-over-18-år-søges-til-projekt-omkring-betydning-af-energitilgængeligheden.aspx